CLINICAL TRIAL: NCT01312740
Title: Effects of Two Hypocaloric Diets on Weight Loss and Inflammatory Markers
Brief Title: Effects of Two Hypocaloric Diets on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceprodi S.A. Kot (Industry)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Pierre and Marie Curie University (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Dr Florence Massiera, Ceprodi S.A. Kot
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: RCB: 2007-A00329-44
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Obesity
Keywords: obesity; dietary treatment; high protein diet; Low glycaemic index; adipocytes; fat mass; systemic inflammatory markers; improvement of complications; effect on weight loss
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Other: LC-P-LGI diet — a hypocaloric diet low in lipids (25%) which is compensated by proteins (35%) with no change in carbohydrate content.
Other: LC-CONV — 4-week CONV period consisted in the subjects' consumption of 1200 Kcal/ day (25% protein, 31% lipids, 44% carbohydrates).

SUMMARY:
The investigators evaluated whether an energy-restricted protein diet with low glycaemic index carbohydrates and soluble fibers (LC-P-LGI) would be more effective than a conventional diet (LC-CONV) on weight-loss and related metabolic variables.

DETAILED DESCRIPTION:
The subjects (9 men and 5 post-menopausal women) were randomly allocated, in a cross-over design, to two periods of 4 weeks of an energy restricted diet of 1200 kcal as either a conventional diet (LC- CONV) or a special energy restricted diet compensated by proteins (LC-P-LGI). The two nutritional periods were separated by a wash-out interval of 8 weeks. Before the start of the study, all subjects were instructed to maintain their usual lifestyle during the experimental period.Anthropometric parameters, glucose and lipid homeostasis and inflammatory markers were evaluated before and after each dietary period.Body fat and fat-free mass distributions were measured by a dual-energy X-ray absorptiometry (DXA, GE Lunar Prodigy Corporation, Madison, WI, USA) before and after each dietary period at the fasting state.

ELIGIBILITY:
Inclusion Criteria:

* BMI 26 to 35 Kg/m2
* 25 to 60 years old
* non diabetic subjects

Exclusion Criteria:

* SGOT and SGPT >2.5x the normal
* plasma glucose more than 1.26 g/l
* hepatic or renal or cardiac failure

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistant pubique-hopitaux Paris, Paris, France

REFERENCES:
- [Derived] Rizkalla SW, Prifti E, Cotillard A, Pelloux V, Rouault C, Allouche R, Laromiguiere M, Kong L, Darakhshan F, Massiera F, Clement K. Differential effects of macronutrient content in 2 energy-restricted diets on cardiovascular risk factors and adipose tissue cell size in moderately obese individuals: a randomized controlled trial. Am J Clin Nutr. 2012 Jan;95(1):49-63. doi: 10.3945/ajcn.111.017277. Epub 2011 Dec 14. PMID 22170375